CLINICAL TRIAL: NCT02406300
Title: Contribution Of Anesthesia Technique For Post-operative Mortality Reduction After Proximal Femur Fractures Surgical Treatment - A Randomized Clinical Trial
Brief Title: Anesthesia And Post-operative Mortality After Proximal Femur Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational changes made recruitment no longer possible
Sponsor: Centro Hospitalar do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); Universidade do Porto (Other)
Responsible Party: Principal Investigator, Raul Carvalho, Raul Carvalho, MD, MSc, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 226-14 (165-DEFI/193-CES)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hip Fractures
Keywords: Hip Fracture; Regional Anesthesia; Peripheral Nerve Blocks; Post-operative Mortality; Cognitive Dysfunction; Quality of Life
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction | interventions — Ropivacaine; Sevoflurane; Desflurane; Bupivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subarachnoid anesthesia (Active Comparator): Patients submitted to subarachnoid anesthesia for proximal femur fracture surgical repair.
  Up to 12.5 mg of bupivacaine or levobupivacaine will be used
  Interventions: Procedure: Subarachnoid Anesthesia; Drug: bupivacaine or levobupivacaine
- PNB/GA (Active Comparator): Patients are submitted to a femoral, a lateral cutaneous nerve of the thigh and an anterior obturator nerve blocks with ropivacaine and an inhalational general anesthesia with sevoflurane or desflurane
  Interventions: Procedure: PNB/GA; Drug: ropivacaine; Drug: sevoflurane or desflurane

INTERVENTIONS:
Procedure: Subarachnoid Anesthesia
  Arms: Subarachnoid anesthesia
Procedure: PNB/GA
  Arms: PNB/GA
Drug: ropivacaine
  Arms: PNB/GA
Drug: sevoflurane or desflurane
  Arms: PNB/GA
Drug: bupivacaine or levobupivacaine
  Arms: Subarachnoid anesthesia

SUMMARY:
This study evaluates the effect of anesthesia on mortality after surgical repair of proximal femur fracture.

Patients will receive either a subarachnoid block or a combination of peripheral nerve blocks and light general anesthesia (PNB/GA).

The investigators hypothesis is that a combination of peripheral nerve blocks with an opioid free light anesthesia may have more favourable outcomes.

Both groups will be followed up for assessment of post-operative morbidity and mortality.

DETAILED DESCRIPTION:
Proximal femur fracture is one of the most common causes of admission in emergency departments. Mortality is high among these patients and is reported to range from 10% at 30 days, up to 32% at one-year post-operative.

Several strategies to reduce mortality have been used, but mortality rate has plateaued since 1998. Attempts to show benefit from regional or general anesthesia have shown inconsistent results. New techniques with peripheral nerve blocks have been used, but their effect on mortality when used as major anesthesia component have not been studied.

The investigators hypothesise that smaller physiologic impact of peripheral nerve blocks associated to light general anesthesia may improve survival rates and reduce short term delirium after proximal femur fracture surgery. Recovery of quality of life will also be assessed.

Patients will be randomized into two groups, being allocated for a subarachnoid anesthesia or a combination of peripheral nerve blocks and light general anesthesia.

Patients will be followed up for short-term post-operative complications such as incidence of delirium, recovery of quality of life and survival up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted wiht a diagnosis of proximal femur fracture (ICD-9 codes 820.0 to 820.9) and submitted to surgical internal fixation of femur or hip prosthesis (ICD-9 codes 7935, 8151 and 8152)

Exclusion Criteria:

* Multiple fractures; polytrauma, active malignancy, ASA(American Society of Anesthesia) status 5, antiplatelet drugs (other than aspirin) in the previous 5 days, known allergies to local anesthetics, contra-indication to general or regional anesthesia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Survival rate | up to one year post-operative

SECONDARY OUTCOMES:
Incidence of post-operative delirium | Up to one week post-operative
  Measured with the 3D-CAM Questionaire (Confusion Assessment Method)
Quality of Life Recovery | Up to one year post-operative
  Quality of Life Assessment tools (SF12v2; EQ-5D (EuroQol); Post-operative Quality Recovery Scale) used from 30 days to one year post-operative. Comparing with pre-surgical values

CONTACTS AND LOCATIONS:
Overall Officials: Raul Carvalho, MSc, Principal Investigator — Serviço de Anestesiologia, Centro Hospitalar do Porto; Faculdade de Medicina, Universidade do Porto; Luís Azevedo, PhD, Study Chair — Universidade do Porto; Fernando Abelha, PhD, Study Chair — Universidade do Porto
Locations (1):
- Serviço de Anestesiologia - Centro Hospitalar do Porto, Porto, Portugal

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043